CLINICAL TRIAL: NCT06969898
Title: Penyagolosa Trail Saludable 2025
Acronym: PTS2025
Status: Completed | Type: Observational
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Other Study IDs: PTS2025 CEISH/103/2024
Record Dates: First submitted 2025-03-17; First posted 2025-05-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Physical Exercise
Keywords: Ultramarathon; biomarkers; Muscle damage; recovery; runners; ultrasound
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Ultramarathon runners: All participants underwent the same protocol: two laboratory assessments, a 106 km race, and post-race physiological parameter evaluations at 24 hours and 48 hours.
  Interventions: Other: Single Ultramarathon runners

INTERVENTIONS:
Other: Single Ultramarathon runners — All participants underwent the same protocol: two laboratory assessments, a 106 km race, and post-race physiological parameter evaluations at 24 hours and 48 hours.

SUMMARY:
The research team leading this project frames it within the objective of advancing knowledge about what happens to this group of athletes who participate in Ultratrail events, with the particularity of studying them during the race itself. To achieve this, the study aims to address four key perspectives.

First, it seeks to understand the training habits of male and female Ultratrail runners. Second, it aims to assess their physical condition and analyze how uphill and downhill segments affect their muscle performance, running efficiency, and strength levels. Third, it investigates the key factors that determine the prediction of race performance for both male and female runners. Finally, the fourth objective is to examine sex differences as a conditioning factor in physiological processes.

DETAILED DESCRIPTION:
There is a category of sporting events held in natural environments over very long distances, classified as Ultratrail races. These races have grown in popularity, attracting an increasing number of participants.

Such races induce states of exhaustion and fatigue, with performance being influenced by numerous factors (environmental conditions, terrain, course profile, etc.), in addition to the athlete's individual characteristics. Scientific interest in these events has surged, and the research community is closely monitoring the health status of participants and their involvement in such races. The aim is to identify the factors influencing performance in a 106 km race (Castelló-Penyagolosa of Penyagolosa Trails) and to assess the physiological impact of participating in this type of endurance event.

To conduct this study, data collection took place before the race, during the race, and within the 48-hour post-race recovery phase.

Before the race, two laboratory sessions were conducted to analyze the athlete's physical condition and assess muscle damage under conditions of both uphill and downhill running. Blood samples were taken before and after these tests.

On race day, measurements included strength loss, weight, dehydration levels, race nutrition, and the evolution of physiological parameters through blood and urine analyses conducted before and after the race.

Finally, blood samples were collected at 24-hours and 48-hours post-race to track the progression of physiological parameters during the recovery phase.

ELIGIBILITY:
Inclusion Criteria:

* Adults healthy with 18-60 years
* Must have completed at least two races of 65 km or longer.
* Must be registered as a participant in the CSP 2025 race

Exclusion Criteria:

* Having heart disease
* Having kidney disease
* Taking a medication on an ongoing basis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ultra-trail runners that will participate in the CSP2025 race (Castellón, Spain; 2025/04/11-12)
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Physiological Parameters | From the enrollment to 48 hours post-race (12 weeks). Baseline (4 weeks after enrollment), post-1-2-3 and 4, 11th week (11 weeks after baseline)
  Blood Analysis: Blood samples will be analyzed for the following parameters:
  * Number of red cells in a volume of blood in µL. (number of red cells x10^6 / µL )
  * Creatine Kinase (CK) in International Units in a volume of blood in litres. (U/L)
  * Lactate Dehydrogenase (LDH) in International Units in a volume of blood in litres. (U/L)
  * C-reactive Protein (CRP) in milligrams in a volume of blood in litres. (mg/L)
  * Sodium (Na) in millimoles in a volume of blood in litres (mmol/L)
  * Potassium (K) in millimoles in a volume of blood in litres (mmol/L)
  * Interleukin 6 (IL-6) in picograms in a volume of blood (pg/dL)
  Blood Sample Collection: Blood samples will be collected twice during the second laboratory session-once before starting the treadmill test (negative 15% incline for 5 km at VT1 speed) and again 30 minutes after completing the test. Additional blood samples will be taken at baseline before the race, at the finish line, 24 hours post-race, and 48 hours post-race.
Muscle Damage | From the enrolment to 48 hours post-race (12 weeks). First measured of knee and ankle extensors will be in 5th week (4 weeks after baseline). Second, and third measured of knee and ankle extensors will be in 11th week (10 weeks after baseline).
  The knee extensors will be measured using ultrasound. Muscle fibre thickness of Rectus femoris and Vastus lateralis will be measured in cm.
  Pennation angle of muscle fibre of Rectus femoris and Vastus lateralis will be measured in degrees.
  The ankle extensors will be measured using ultrasound. Muscle fibre thickness of Medial gastrocnemius will be measured in cm. Pennation angle of muscle fibre of Medial gastrocnemius will be measured in degrees.
  Assessments will be conducted twice during the second laboratory session: once before starting the treadmill test (-15% incline for 5 km at VT1 speed) and again 30 minutes after completing the test. Additionally, measurements will be taken at baseline before the race start and at the finish line
Strength levels | First SJ measured (first week), second SJ at day before the race (11th week) third SJ at the end of the race (11th week). RSI will be measured at the first laboratory session (1st week). MIS will be measured at the second laboratory session (5th week)
  Measurements:
  * Squat Jump (SJ): Jump height in centimetres will be measured during a vertical jump performed from a squat position without a countermovement.
  * Reactive Strength Index (RSI): The subject performs a sequence of 10 consecutive jumps, during which flight time (in milliseconds) and ground contact time (in milliseconds) are measured. These two variables are used to calculate the Reactive Strength Index (RSI), defined as the ratio of flight time to contact time (flight time in milliseconds / contact time in milliseconds).
  * Maximal Isometric Strength (MIS): The isometric strength of the knee and ankle extensors will be measured in Newtons (N).
  Collection of Measurements: • Squat Jump will be evaluated during the first laboratory session (first week), before and after cardiopulmonary test (two jumps per attempt). • Reactive Jump will be assessed during the first laboratory session (first week), before and after the 5 km at VT1 speed treadmill test (-15% incline)
Physical activity data | Laboratory 4 weeks before the race. During the race 96 hours (from the day before the race to 48hours post-race)
  Accelerometry:
  Physical activity (counts per minute, CPM) will be measured using an accelerometer placed on the non-dominant wrist. Activity levels will be classified into six categories: sedentary, light, moderate, vigorous, very vigorous, and extremely vigorous.
  Collection of Measurements:
  * Accelerometry will be recorded during laboratory assessments.
  * An accelerometer will be placed on the participant the day before the race to continuously collect physical activity data until 48 hours post-race.
Physiological Parameters | At the start line of the race (11th week) and at the end of the race (11th week)
  Urine Samples:
  Urinary density (mg/dL)
  Urine samples will be collected at baseline before the race and at the finish line, with measurements of urinary density (Units: mg/dL).

SECONDARY OUTCOMES:
Body Composition & Anthropometry | Baseline (1st week)
  Weight in kilograms, height in meters. Weight and height will be combined to report BMI in kg/m^2.
  Assessed using bioelectrical impedance analysis (BIA) to estimate percentage of fat mass (%), percentage of fat-free mass (%), and total body water (L). The percentage of fat mass (%), percentage of fat-free mass (%), and total body water (L) will be used to know the body composition of the subject combining the percentage of fat mass, percentage of fat free mass and total body water.
  Collection of Measurements:
  • Weight, height, BMI, percentage of fat mass, percentage of fat-free mass, total body water and Body composition will be measured during the first laboratory assessment (1st week)
Physical Condition | Baseline (1st week) and post baseline (5th week)
  Maximal Oxygen Consumption (V ̇O2max):
  Number of millilitres of oxygen consumption, weight in kilograms and time in minutes will be combined to calculated the Maximal Oxygen Consumption. Millilitres per kilogram per minute (mL/kg/min).
  Oxidation Substrate Levels: Assessed through indirect calorimetry to determine number of carbohydrate grams and number of fat grams oxidation rates per minute (g/min).
  Collection of Measurements:
  * V ̇O2max will be evaluated in baseline laboratory assessment (1st week).
  * Oxidation substrate levels will be measured during the second laboratory assessment (5th week).
Muscle Oxygenation Measurement | Baseline (Day 1) and post baseline (4 weeks after baseline)
  Oxygen Saturation Levels: Measured in the muscles involved in running using near-infrared spectroscopy (NIRS) and expressed as a percentage (%).
  Collection of Measurements: Oxygen saturation levels will be assessed during two laboratory tests.
Running Power Measurement | Baseline (Day 1) and post baseline (4 weeks after baseline)
  Power Output: Measured in watts (W) using a power meter to assess mechanical performance during running.
  Collection of Measurements: Power output will be recorded during the two treadmill tests conducted in the laboratory.
Weight | The start line of the race (11th week), during the intervention three times during the race (in km 32, in km 62 and in km 81) and at the end of the race (11th week)
  Body mass (kg)
  Weight is measured in kilograms at the starting line, at three race checkpoints (32 km, 62 km, and 81 km), and at the finish line.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hernando, Principal Investigator — Universitat Jaume I
Locations (1):
- Jaume I Univesity, Castellon, Castellón, Spain

REFERENCES:
- [Background] Hernando C, Hernando C, Collado EJ, Panizo N, Martinez-Navarro I, Hernando B. Establishing cut-points for physical activity classification using triaxial accelerometer in middle-aged recreational marathoners. PLoS One. 2018 Aug 29;13(8):e0202815. doi: 10.1371/journal.pone.0202815. eCollection 2018. PMID 30157271
- [Background] Guerrero C, Collado-Boira E, Martinez-Navarro I, Hernando B, Hernando C, Balino P, Muriach M. Impact of Plasma Oxidative Stress Markers on Post-race Recovery in Ultramarathon Runners: A Sex and Age Perspective Overview. Antioxidants (Basel). 2021 Feb 27;10(3):355. doi: 10.3390/antiox10030355. PMID 33673404
- [Background] Granero-Gallegos A, Gonzalez-Quilez A, Plews D, Carrasco-Poyatos M. HRV-Based Training for Improving VO2max in Endurance Athletes. A Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2020 Oct 30;17(21):7999. doi: 10.3390/ijerph17217999. PMID 33143175
- [Background] Baygutalp F, Buzdagli Y, Ozan M, Koz M, Kilic Baygutalp N, Atasever G. Impacts of different intensities of exercise on inflammation and hypoxia markers in low altitude. BMC Sports Sci Med Rehabil. 2021 Nov 22;13(1):145. doi: 10.1186/s13102-021-00375-0. PMID 34809670
- [Background] Baird MF, Graham SM, Baker JS, Bickerstaff GF. Creatine-kinase- and exercise-related muscle damage implications for muscle performance and recovery. J Nutr Metab. 2012;2012:960363. doi: 10.1155/2012/960363. Epub 2012 Jan 11. PMID 22288008